CLINICAL TRIAL: NCT01025193
Title: One Year Exploratory Study to Evaluate the Efficacy and Safety of Belimumab for Normalization of Alloantibody Levels in Sensitized Patients Awaiting Kidney Transplantation
Brief Title: Desensitization With Belimumab in Sensitized Patients Awaiting Kidney Transplant
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: has not demonstrated efficacy in primary goal
Sponsor: University of Pennsylvania (Other)
Collaborators: Human Genome Sciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IND 106342
Record Dates: First submitted 2009-12-01; First posted 2009-12-03 (Estimated); Results first posted 2017-02-28 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-05

CONDITIONS: Desensitization
Keywords: belimumab; Benlysta; LymphoStat B; BLyS specific inhibitors
MeSH Terms: interventions — belimumab

STUDY DESIGN:
Intervention Model Description: There was only one group in this trial. All participants received belimumab.
Masking Description: There was no masking in this single group trial. The patients, providers and investigators were all aware that the patient were on belimumab therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Belimumab (Experimental): Belimumab will be administered intravenously at a dose of 10mg/kg on days 0, 14, 28 and every 28 days for up to 52 weeks to normalize alloantibody levels in sensitized patients awaiting kidney transplantation. Subjects who are not able to undergo transplantation before the end of the treatment period will have final follow-up evaluation 8 weeks after the last dose of belimumab is administered.
  Interventions: Drug: Belimumab

INTERVENTIONS:
Drug: Belimumab — Belimumab is a fully human monoclonal antibody that recognizes and inhibits BLyS ®. BLyS ® is a B-lymphocyte stimulator protein which plays a role in the development of B lymphocyte cells into plasma B cells, which then produce antibodies that can sensitize a potential transplant recipient. At the time of this trial, belimumab was not yet FDA approved and was being studied in clinical trials for the treatment of systemic lupus erythematosus. Until this trial, it had not yet been used in the transplant setting.
  Other Names: registered name Benlysta; also previously known as LymphoStat-B

SUMMARY:
If subjects are listed for kidney transplant and are considered sensitized, this means they have a high amount of antibodies in their blood that could react to a kidney transplant offered for them. Antibodies are protein substances made by the body that fight anything that the body considers as a threat to it, such as infection or a kidney transplant. Sensitization may be due to prior transplants, pregnancy, or blood transfusions. Being sensitized can increase the subject's kidney transplant waiting time as it is more difficult to find a suitable kidney transplant for them that their antibodies will not react to. The purpose of this research study is to see if giving the investigational drug belimumab up to one year pre-transplant can de-sensitize the subjects, or decrease the amount of antibodies in their blood. This may help make the subjects eligible to receive a kidney transplant more quickly. If after receiving belimumab, the subjects are compatible with a donor kidney offered and are medically suitable for transplant at that time, a kidney transplant will be performed.

DETAILED DESCRIPTION:
Approximately one third of patients awaiting kidney transplant at our transplant center have significant levels of antibodies in their blood leading to a longer wait time for a kidney transplant and death. Antibodies in the blood may be due to prior transplants, pregnancy, or blood transfusions. These antibodies sensitize a patient and make it more difficult for the patient to get a compatible kidney transplant. The measure of these antibodies is called panel reactive antibodies (PRA) and can range from 0-100%, with 100% being most sensitized. The waiting time for patients with a PRA in the range of 20%-79% is over 5 years as compared to patients with low PRA (0%-19%) which is 3-4 years. Patients with a PRA greater than 80% are likely to be granted extra points to increase the chances of transplantation. Antibodies in these patients may be due to prior transplants, pregnancy, or blood transfusions. To date, no trials with belimumab have been performed in patients with pre-existing antibodies awaiting kidney transplantation. This study is undertaken to assess the effectiveness and safety of using belimumab to normalize antibody levels in sensitized patients awaiting kidney transplantation. It is hoped that decreasing these antibodies will decrease the waiting time on the kidney transplant list, and allow the patient to become compatible with a donor kidney for transplant.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 -75 years.
* Patients denied a kidney transplant because of a prior positive crossmatch
* Patients awaiting a first or second kidney transplant from a living or deceased donor
* Patients who have given written informed consent to participate in all aspects of the study.
* Patients with no potential living donors should have accumulated at least 12 months waiting time in our organ procurement organization
* And one of the following criteria:
* Pre-sensitized patients defined by Luminex antibody assays and whose panel reactive antibody (PRA) is 20% or greater
* Patients with a PRA of less than 20% but who have HLA antibody specificities to HLA-Cw, DP or allele-specific antigens

Exclusion Criteria:

* Patients with known hypersensitivity to belimumab or who have received biologics, within the last 90 days
* Patients receiving corticosteroids, intravenous immunoglobulin, cyclophosphamide, mycophenolate mofetil, or azathioprine from 90 days prior to study entry until day of transplant.
* Patients with a history of anaphylaxis to parenteral administration of contrast agents, foreign proteins, or monoclonal antibodies.
* Patients with multi-organ transplant
* Patients who have received any investigational immunosuppressive drug within 1 month of inclusion into this study or if use of such a product is anticipated.
* Patients who have received any live vaccine within 30 days of study entry.
* Female patients who are pregnant, lactating.
* Female patients of child bearing potential and not willing to practice an approved method of birth control for 1 month prior to the start of the study agent and 8 weeks after the last dose of study agent.
* Male patients who are not agreeable to using effective contraception throughout the study and for 3 months after the last dose of study agent.
* Patients with a known malignancy or history of malignancy other than excised basal or squamous cell carcinoma of the skin.
* Patients who are positive for Hepatitis B infection, Hepatitis C infection or Human Immunodeficiency Virus (HIV)-positive patients.
* Patients with evidence of severe liver disease, including abnormal liver profile tests > 3 times upper limit of normal at screening.
* Patients with current severe infection.
* Patients with any surgical or medical condition, which in the opinion of the investigator precludes enrollment in this trial
* Patients who live far from the transplant center and are unable to comply with all study visits.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-02; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ali Naji, MD, Ph D, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsyvlania Kidney Transplant Program, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From April 2010 to October 2011 patients listed for renal transplant at the Hospital of the University of Pennsylvania who met study inclusion criteria and none of the exclusion criteria were approached during an outpatient clinic visit to participate in the study.
Pre-assignment Details: There were no wash out, run-in or transition periods for this trial.
Groups:
- Belimumab: Belimumab is a monoclonal antibody. It is the first drug of its type in a new class of medications called BLyS-specific inhibitors. In March 2011, it was approved by the Food and Drug Administration (FDA) for the treatment of adult patients with active, autoantibody-positive, systemic lupus erythematosus (SLE) who are receiving standard therapy. In this study, belimumab was being used to try to decrease the amount of antibodies in the subject's blood pre-kidney transplant. This use was considered investigational (not approved by the Food and Drug Administration).
  Belimumab : The subjects were given this medication as an outpatient as an intravenous infusion through the arm. The medication was given at the beginning of the study, two weeks later, and then every 4 weeks for up to one year pre-transplant.
Period: Overall Study
Arm/Group | Belimumab
Started | 8
Completed | 4 (one patient was transplanted 2 weeks after 8 month belimumab dose and did not receive further doses.)
Not Completed | 4
Not completed — Protocol Violation | 1
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Groups:
- Belimumab: Belimumab is a monoclonal antibody. It is the first drug of its type in a new class of medications called BLyS-specific inhibitors. In March 2011, it was approved by the Food and Drug Administration (FDA) for the treatment of adult patients with active, autoantibody-positive, systemic lupus erythematosus (SLE) who are receiving standard therapy. In this study, belimumab was used in to try to decrease the amount of antibodies in the pre-kidney transplant patient's blood. This use was considered investigational (not approved by the Food and Drug Administration).
  Belimumab : The subjects were given this medication as an outpatient as an intravenous infusion through the arm. The medication was given at the beginning of the study, two weeks later, and then every 4 weeks for up to one year pre-transplant.
Arm/Group | Belimumab
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness of Belimumab to Normalize Allo-antibody Levels in Sensitized Patients Awaiting Kidney Transplantation.
Description: Before transplant it is necessary to measure antibodies that the recipient might have and compare them to the living or decease donor's immune make-up. Recipients with many antibodies or a specific antibody in a high concentration may have a more difficult time finding a compatible donor, and being transplanted. These recipients are referred to as sensitized patients. It is important that the sensitized recipient and the donor be compatible to prevent rejection after transplant. We measured antibodies levels in sensitized patients waiting for kidney transplant, to see if belimumab would decrease these antibody levels.
Time Frame: up to one year pre-transplant
Population: any patient who received at least one dose of belimumab was included in analysis population
Measure: Count of Participants; unit: Participants
Arm/Group | Belimumab
Number analyzed (Participants) | 8
Participants
  Patients not experiencing a decrease in antibodies | 8
  Patients experiencing a decrease in antibodies | 0

2. Primary Outcome: Successful Kidney Transplantation From a Cross-match Compatible Donor (as a Result of Belimumab Therapy)
Description: In order for a sensitized recipient ( a recipient with antibodies) to be transplanted, the cross match with the donor has to be compatible. We wanted to study if belimumab reduced antibodies in sensitized patients and led those patients to subsequently become cross-match compatible with a donor and allow for successful transplant.
Time Frame: one year pre-transplant
Population: All participants enrolled who received at least one dose of belimumab were considered for analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Belimumab: Belimumab is a monoclonal antibody. It is the first drug of its type in a new class of medications called BLyS-specific inhibitors. In March 2011, it was approved by the Food and Drug Administration (FDA) for the treatment of adult patients with active, autoantibody-positive, systemic lupus erythematosus (SLE) who are receiving standard therapy. In this study, belimumab is being used in to try to decrease the amount of antibodies in the subject's blood pre-kidney transplant. This use is considered investigational (not approved by the Food and Drug Administration).
  Belimumab : The subjects will be given this medication as an outpatient as an intravenous infusion through the arm. The medication will be given at the beginning of the study, two weeks later, and then every 4 weeks for up to one year pre-transplant.
Arm/Group | Belimumab
Number analyzed (Participants) | 8
Participants
  Kidney transplant as a result of belimumab therapy | 0
  kidney transplant unrelated to belimumab therapy | 1
  Kidney transplant not received during trial | 7

3. Secondary Outcome: Pharmacokinetics of Belimumab Measured as Number of Participants With Specific Dilution Factors at Each Time Point.
Description: We wanted to look at belimumab pharmacokinetics in sensitized patients awaiting kidney transplant. These are reported as number of participants with specific dilution factors at each studied time-point. Blood for these tests could be drawn pre dose as well as 0-4 hours after the dose was given. Belimumab dilutions factors were measured pre dose at timepoints 0 (first day of belimumab), days 56 and 364. Belimumab dilution factors were measured after the dose on days 14, and 168. Belimumab dilution factors were also measured at 8 weeks after completion of belimumab therapy and pre dose at any unscheduled visits if needed.
Time Frame: Belimumab serum drug dilution factors were measured in patients at at timepoints 0 (first day of belimumab), day 14, day 56, day 168, 364, at any unscheduled visits, and at 8 weeks post completion of belimumab therapy.
Population: any patient who received at least one dose of belimumab was included in the analysis
Measure: Count of Participants; unit: Participants
Groups:
- Belimumab: Belimumab is a monoclonal antibody. It is the first drug of its type in a new class of medications called BLyS-specific inhibitors. In March 2011, it was approved by the Food and Drug Administration (FDA) for the treatment of adult patients with active, autoantibody-positive, systemic lupus erythematosus (SLE) who are receiving standard therapy. In this study, belimumab was used to try to decrease the amount of antibodies in the pre-kidney transplant patient's blood. This use was considered investigational (not approved by the Food and Drug Administration).
  Belimumab : The subjects were given this medication as an outpatient as an intravenous infusion through the arm. The medication was given at the beginning of the study, two weeks later, and then every 4 weeks for up to one year pre-transplant.
Arm/Group | Belimumab
Number analyzed (Participants) | 8
Participants
  Pre Dose Belimumab Serum Dilution at 400-Day 0 | 8
  Pre Dose Belimumab Serum Dilution at 8000-Day 56: number analyzed (Participants) | 7
  Pre Dose Belimumab Serum Dilution at 8000-Day 56 | 7
  Pre Dose Belimumab Dilution 8000 at Day 364: number analyzed (Participants) | 2
  Pre Dose Belimumab Dilution 8000 at Day 364 | 2
  Post Dose Belimumab Dilution at 8000 at Day 14: number analyzed (Participants) | 7
  Post Dose Belimumab Dilution at 8000 at Day 14 | 7
  Post Dose Belimumab Dilution at 8000 at Day 168: number analyzed (Participants) | 6
  Post Dose Belimumab Dilution at 8000 at Day 168 | 6
  Belimumab Dilution 8000 at 8 weeks After Belimumab: number analyzed (Participants) | 2
  Belimumab Dilution 8000 at 8 weeks After Belimumab | 2

4. Secondary Outcome: B and T Lymphocyte Subsets
Description: B and T Lymphocyte subsets were measured through flow cytometry pre-treatment and at months 1,2,12 and at 8 weeks after the last belimumab dose. We looked for clinically significant changes (as determined by Principal Investigator) in these subsets at each time-point.
Time Frame: 8 weeks after the last dose of belimumab
Population: Any patient who received at least one dose of belimumab was included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Belimumab
Number analyzed (Participants) | 8
Participants
  Decrease in T and B Cell Flow Cytometry:month 1: number analyzed (Participants) | 7
  Decrease in T and B Cell Flow Cytometry:month 1 | 0
  Decease in T and B Cell Flow Cytometry:month 2: number analyzed (Participants) | 7
  Decease in T and B Cell Flow Cytometry:month 2 | 0
  Decrease in T and B Cell Flow Cytometry:month 12: number analyzed (Participants) | 3
  Decrease in T and B Cell Flow Cytometry:month 12 | 0
  Decrease in T and B Cell Flow Cytometry:post 8 wks: number analyzed (Participants) | 3
  Decrease in T and B Cell Flow Cytometry:post 8 wks | 0

5. Secondary Outcome: BLyS Levels Before and After Treatment With Belimumab
Description: We assessed for unexpected changes in bound and unbound BLyS levels before and after treatment with belimumab. These were measured from before treatment and at months 1,2,6,10 and 12 months after belimumab treatment and again at 8 weeks after belimumab treatment.
Time Frame: up to 8 weeks after completion of therapy
Population: Any patient who received at least one dose of belimumab was included in the analysis
Measure: Count of Participants; unit: Participants
Groups:
- Belimumab: Belimumab is a monoclonal antibody. It is the first drug of its type in a new class of medications called BLyS-specific inhibitors. In March 2011, it was approved by the Food and Drug Administration (FDA) for the treatment of adult patients with active, autoantibody-positive, systemic lupus erythematosus (SLE) who are receiving standard therapy. In this study, belimumab is being used in to try to decrease the amount of antibodies in the subject's blood pre-kidney transplant. This use is considered investigational (not approved by the Food and Drug Administration).
  Belimumab: The subjects will be given this medication as an outpatient as an intravenous infusion through the arm. The medication will be given at the beginning of the study, two weeks later, and then every 4 weeks for up to one year pre-transplant.
Arm/Group | Belimumab
Number analyzed (Participants) | 8
Participants
  Unexpected change in BLyS levels at 1 month: number analyzed (Participants) | 7
  Unexpected change in BLyS levels at 1 month | 0
  Unexpected change in BLyS levels at 2 month: number analyzed (Participants) | 7
  Unexpected change in BLyS levels at 2 month | 0
  Unexpected change in BLyS levels at 6 mo: number analyzed (Participants) | 6
  Unexpected change in BLyS levels at 6 mo | 0
  Unexpected change in BLyS levels at 12 months: number analyzed (Participants) | 3
  Unexpected change in BLyS levels at 12 months | 0
  Unexpected change in BLyS levels 8 wks post treat: number analyzed (Participants) | 3
  Unexpected change in BLyS levels 8 wks post treat | 0

6. Secondary Outcome: Hepatitis B Vaccine Antibody Titers
Description: We investigated if belimumab treatment would decrease Hepatitis B vaccine titers by 12 months after treatment with belimumab. All patients received Hepatitis B vaccine before beginning treatment with belimumab.
Time Frame: up to 12 months of treatment with belimumab
Population: All patients who received at least one dose of belimumab were included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Belimumab
Number analyzed (Participants) | 7
Participants
  Patients who maintained Hepatitis B titer | 7
  Patients who did not maintain Hepatitis B titer | 0

7. Secondary Outcome: Number of Participants With Treatment Related Serious Adverse Events
Description: To assess the safety of belimumab in sensitized patients awaiting kidney transplant we evaluated the number of participants with serious adverse events possibly or definitely related to belimumab.
Time Frame: up to one year pre-transplant
Population: Any patient who received at least one dose of belimumab was included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Belimumab
Number analyzed (Participants) | 8
Participants
  Hives/infusion reaction related to belimumab | 1
  No SAEs possibly/definitely related to belimumab | 7

ADVERSE EVENTS:
Time Frame: adverse events were collected for up to 12 months during which patients received belimumab therapy and for 8 weeks after the last dose of belimumab therapy.
Groups:
- Belimumab: Belimumab is a monoclonal antibody. It is the first drug of its type in a new class of medications called BLyS-specific inhibitors. In March 2011, it was approved by the Food and Drug Administration (FDA) for the treatment of adult patients with active, autoantibody-positive, systemic lupus erythematosus (SLE) who are receiving standard therapy. In this study, belimumab was used to try to decrease the amount of antibodies in the patient waiting for kidney transplant's blood. This use was considered investigational (not approved by the Food and Drug Administration).
  Belimumab : The subjects were given this medication as an outpatient as an intravenous infusion through the arm. The medication was given at the beginning of the study, two weeks later, and then every 4 weeks for up to one year pre-transplant.
Arm/Group | Belimumab
Serious Adverse Events (participants affected / at risk) | 3/8
Other Adverse Events (participants affected / at risk) | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belimumab (N=8)
Atrial Fibrillation (Cardiac disorders) | 1 (1) — unrelated to study drug
Atrial Ablation (Cardiac disorders) | 1 (1) — unrelated to study drug
Anemia (Blood and lymphatic system disorders) | 1 (1) — unrelated to study drug, occurred post-transplant in 8 week belimumab follow-up phase
fluid overload (Renal and urinary disorders) | 1 (1) — unrelated to study drug in both cases, occurred post-transplant in 8 week post belimumab follow-up phase in 1 patient
hives (Immune system disorders) | 1 (1) — related to study drug at first dose
Infusion reaction (Injury, poisoning and procedural complications) | 1 (1) — allergic reaction to first dose of study drug
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belimumab (N=8)
Rash left antecubitus from adhesive tape (Skin and subcutaneous tissue disorders) | 1 (1) — unrelated to study drug
Hypertensive episode (Renal and urinary disorders) | 1 (1) — unrelated to study drug
Electrolyte imbalance (Renal and urinary disorders) | 1 (1) — unrelated to study drug
Nausea (Gastrointestinal disorders) | 1 (1) — related to menstrual cycle per patient, unrelated to study drug
non-cardiac related chest pain (General disorders) | 1 (1) — non cardiac related, resolved on own, unrelated to study drug
Shakiness (General disorders) | 1 (1) — patient seen in ER, but no cause identified and resolved, unrelated to study drug
anemia (low red blood cell count) (Blood and lymphatic system disorders) | 1 (1) — unrelated to study drug, continued from SAE, post renal transplant
fluid overload (Renal and urinary disorders) | 1 (2) — not related to study drug
infection cold symptoms (Infections and infestations) | 1 (1) — unrelated to study drug
partial parathyroidectomy (Endocrine disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Few patients enrolled, and limited follow-up due to trial being halted due to lack of efficacy after review by investigators and the data safety monitoring board. Only one patient was transplanted during the trial (unrelated to study treatment).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No